CLINICAL TRIAL: NCT02594566
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Prophylactic Cytomegalovirus Plasmid DNA Vaccine in Healthy Adults
Brief Title: Safety, Tolerability, and Immunogenicity of a Cytomegalovirus DNA Vaccine
Acronym: CM04-101
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Vical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HM20004886
Record Dates: First submitted 2015-10-16; First posted 2015-11-03 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Cytomegalovirus; Vaccine; Congenital Infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — vaxfectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research Subjects (Experimental): A total of 3 injections of the vaccine (CyMVectin) will be given at Days 0, 28 (+4 days), and 56 (+4 days).
  Interventions: Drug: CyMVectin

INTERVENTIONS:
Drug: CyMVectin — CyMVectin will be delivered by unilateral intramuscular (IM) injection at Day 0, Day 28(+4 days), and Day 56 (+4 days) in alternating arms. Each dose of CyMVectin will be administered in a 1.0-mL volume
  Other Names: VCL-6365; Vaxfectin

SUMMARY:
If the participant decides to take part in the study, the participant will need to do the following:

Visit the study clinic up to 10 times and be available for a reasonable amount of follow up phone calls to see how the participant is doing.

The participant will receive three doses of vaccine injected into the muscle of the upper arm. After each injection the participant will be asked to remain at the study site for at least 30 minutes after the participant receives the study vaccine.

The results of all of the participants blood tests, just like all other laboratory test results, will be provided to the Investigators, Sponsor, and vaccine developer. Positive HIV and viral hepatitis test results will be reportable to local health authorities according to local laws.

The participant will be asked to refrain from excessive physical activities and alcohol consumption within 2 days before each clinic visit to avoid possible confusing effects on laboratory tests.

DETAILED DESCRIPTION:
Up to 10 normal healthy adult female subjects 18 to 35 years of age will be enrolled in this trial. A total of 3 injections of the vaccine will be given at Days 0, 28 (+4 days), and 56 (+4 days). There are follow-up visits 7 days after each vaccination, one follow-up visit 28 days after the 3rd (last) vaccination, and a final visit 3 months later. Blood and urine samples will be collected at each vaccination and follow-up visit. The participant will be asked to complete a telephone call follow-up at 1 year after receiving the last vaccination.

Participants will be required to complete subject diary cards throughout the study until the telephone call follow-up at approximately Day 420 (i.e., 12 months following the 3rd and final dose scheduled for Day 56). Diary cards will be reviewed with the study staff at each visit and during the Day 420 telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female adults, 18 to 35 years of age
* Able and willing to be followed for approximately 15 months
* Lack serum antibodies specific for CMV
* Able to provide informed consent

Exclusion Criteria:

* History of receiving any previous CMV vaccine
* Pregnant, trying to become pregnant, or breastfeeding
* Receipt or donation of blood, blood products, or plasma within 30 days of the initial injection
* Clinically significant findings from clinical evaluation or laboratory tests, evidence of medical disease(s) or medical/psychiatric condition(s), or unable to participate due to occupation or other social reasons
* Use of immunomodulatory therapy (drugs that suppress the immune system) within the past 6 months or other medications or nutritional supplements as determined by the study investigators that may interfere with the vaccine response, or increase safety risks to the participant, that have been taken within 30 days prior to the initial injection on Day 0
* Antinuclear antibody (ANA) titer >1:80
* Body mass index (BMI) >30
* Less than 18 years of age or older than 35 years of age
* No access to a telephone

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Up to Day 182
Number of participants with treatment-related adverse events of special interest | Up to Day 420

SECONDARY OUTCOMES:
CMV gB antibody and CMV neutralizing antibody responses change from baseline | Baseline, Days 28, 35, 56, 63, 86, 182

CONTACTS AND LOCATIONS:
Overall Officials: Michael A McVoy, Ph.D., Principal Investigator — Virginia Commonwealth University